CLINICAL TRIAL: NCT04389580
Title: Combination Therapy With Isotretinoin and Tamoxifen Expected to Provide Complete Protection Against Severe Acute Respiratory Syndrome Coronavirus
Acronym: Combination
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COV-19 Treatment This is
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Isotretinoin; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 13 cis retinoic acid doses orally plus Tamoxifen orally (Active Comparator): 80 infected patients will receive tamoxifen 20 mg orally twice daily with a glass of water and after three days of the standard therapy the infected patients will receive 13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days
  Interventions: Drug: Drug: Isotretinoin plus Tamoxifen
- 13 cis retinoic acid doses Aerosolized plus Tamoxifen orally (Active Comparator): 80 infected patients will receive tamoxifen 20 mg orally twice daily with a glass of water and after three days of tamoxifen therapy the infected patients will receive Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Interventions: Drug: Aerosolized Isotretinoin plus Tamoxifen
- No Intervention: (No Intervention): No study treatment Arm No Isotretinoin or Tamoxofien treatment

INTERVENTIONS:
Drug: Drug: Isotretinoin plus Tamoxifen — 20 mg PO (by mouth) twice daily for 14 days
  13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days starting after three days of taking tamoxifen
  Arms: 13 cis retinoic acid doses orally plus Tamoxifen orally
Drug: Aerosolized Isotretinoin plus Tamoxifen — 20 mg PO (by mouth) twice daily for 14 days
  Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days starting after three days of taking tamoxifen
  Arms: 13 cis retinoic acid doses Aerosolized plus Tamoxifen orally

SUMMARY:
Combination Therapy with Isotretinoin and Tamoxifen expected to provide Complete Protection against Severe Acute Respiratory Syndrome Coronavirus

Abstract:

The COVID-19 pandemic caused by SARS-COV-2 has infected over 2,000,000 people causing over 150,000 deaths.Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 and for which there are currently no approved treatments.The principal investigator reported according to previous research data that combination therapy with Isotretinoin and tamoxifen expected to provide Complete Protection against Severe Acute Respiratory Syndrome Coronavirus, ACE2-expressing cells can act as home cells and are prone to SARS-CoV-2 infection as ACE2 receptor facilitates cellular viral entry and replication. A study demonestrated that patients with hypertension and diabetes mellitus may be at higher risk of SARS-CoV-2 infection, as these patients are often treated with ACE inhibitors (ACEIs) or angiotensin II type-I receptor blockers (ARBs), which have been previously suggested to increase ACE2 expression, In another study by Sinha et al who analyzed a publicly available Connectivity Map (CMAP) dataset of pre/post transcriptomic profiles for drug treatment in cell lines for over 20,000 small molecules, isotretinoin was the strongest down-regulator of ACE 2 receptors. On the other hand, they found 6 drugs in CMAP that are currently being investigated in clinical trials for treating COVID-19 (chloroquine, thalidomide, methylprednisolone, losartan, lopinavir and ritonavir, from clinicaltrials.gov), none of which was found to significantly alter ACE2 expression (P>0.1) Moreover, another study demonstrated that isotretinoin is a Potential papain like protease (PLpro) inhibitors which is a protein encoded by SARS-CoV-2 genes and considered one of the proteins that should be targeted in COVID-19 treatment by performing target-based virtual ligand screening. As Investigators discussed before in their previous clinical trial (NCT04353180) that Isotretinoin is the strongest down-regulator of ACE2. and the principal investigator expects that Isotretinoin can inhibit or downrgulat ACE2 by direct interaction and binding with the transmembrane ACE2, Suggesting its therapeutic potential in preventing the entry of COVID 2019 to the host cell. The second combined drug is tamoxifen, A study demonstrated that tamoxifen causes redistribution of weak base chemotherapeutics from acidic organelles to the nucleus in drug-resistant cells. Agents that disrupt organelle acidification (e.g., monensin, bafilomycin A1) cause a similar redistribution. Measurement of cellular pH in several cell lines reveals that tamoxifen inhibits acidification of endosomes and lysosomes without affecting cytoplasmic pH, Tamoxifen decreased the rate of vesicular transport though the recycling and secretory pathways. Organellar acidification is required for many cellular functions, and its disruption could account for many of the side effects of tamoxifen. A sudy demonstrated that the phagocytosis is inhabited by tamoxifen and chloroquine in retinal epithelial cells and Also, a study demonstrated that Tamoxifen have weak base property and increase endolysosomal pH and alter endosomal dynamics. Importantly, TAM treatment enhanced survival of mice injected with a lethal dose of STx1 or STx2, TAM allowed TAM to increase endolysosomal pH and alter endosomal dynamics. A study demonstrated that Tamoxifen have antimalarial effect via treating mice infected with P. berghei, which show lower levels of parasitaemia and do not develop signs of cerebral malaria, Tamoxifen is found to prevent lung fibrosis and reduce serum TGFβ-1 levels. A study Reported that Tamoxifen have endosomal and lysosomal cysteine proteases inhibitory effect better than chloroquine , Cathepsins are endosomal and lysosomal cysteine proteases that play important roles in protein degradation in various cellular processes including both the endocytic pathway and autophagy. The role of cathepsins in viral infection was first identified by Huang et al and they found that one cysteine proteases inhibitor E64d and a specific cathepsin L inhibitor Z-FY(t-Bu)-DMK are able to block the SARS-CoV infection. A study demonestrated that Cathepsin D was more sensitive to tamoxifen than to chloroquine. Tamoxifen exposures decreased the cathepsin D activity at less than 10 pM concentrations. The effect of chloroquine started at concentration of 15 pM, Finally, the principal investigator expects strong inhibition of COVID-19 by this combination therapy.

In addition, Tamoxifen has anti estrogenic effect Therefore the principal investigator expects that Tamoxifen will protect patients with cancer against COVID-19 infection.

Keywords: COVID 2019 , Isotretinoin , Tamoxofin, ACE2,.Endosomal and Lysosomal pH.

DETAILED DESCRIPTION:
The study is a randomized interventional comparative Phase II trial. The duration of the trial for each subject is expected to be 3 months.160 adult male and female patients with positive COVID-19 diagnosis and fulfilling the below outlined inclusion criteria will be enrolled into the study. Trial population will consist of both genders.

Study Type:Interventional [Change...]

Primary Purpose:Treatment

Study Phase:Phase 2 Interventional Study Model:Sequential Assignment

Number of Arms:3

Masking: None (Open Label)

Allocation:Randomized

Enrollment:160 [Anticipated]

Isotretinoin(13cis RA) may be able to inhibit COVID 2019 entry via down regulation of ACE2 , AT1 protein and Ang II-mediated intracellular calcium release rather than inhibition of interleukin-6 (IL-6) and this is discussed as follow :

The COVID-19 pandemic caused by SARS-COV-2 has infected over 2,000,000 people causing over 150,000 deaths. A key host cellular protein required for the virus entry is angiotensin-converting enzyme 2 (ACE2) whose expression has been demonstrated in many tissues including alveolar epithelial type II cells in lungs, oral mucosa and intestine, heart, kidney, endothelium and skin. ACE2-expressing cells can act as home cells and are prone to SARS-CoV-2 infection as ACE2 receptor facilitates cellular viral entry and replication. A study demonestrated that patients with hypertension and diabetes mellitus may be at higher risk of SARS-CoV-2 infection, as these patients are often treated with ACE inhibitors (ACEIs) or angiotensin II type-I receptor blockers (ARBs), which have been previously suggested to increase ACE2 expression. In another study by Sinha et al who analyzed a publicly available Connectivity Map (CMAP) dataset of pre/post transcriptomic profiles for drug treatment in cell lines for over 20,000 small molecules, isotretinoin was the strongest down-regulator of ACE 2 receptors. On the other hand, they found 6 drugs in CMAP that are currently being investigated in clinical trials for treating COVID-19 (chloroquine, thalidomide, methylprednisolone, losartan, lopinavir and ritonavir, from clinicaltrials.gov), none of which was found to significantly alter ACE2 expression (P>0.1) Moreover, another study demonstrated that isotretinoin is a Potential papain like protease (PLpro) inhibitors which is a protein encoded by SARS-CoV-2 genes and considered one of the proteins that should be targeted in COVID-19 treatment by performing target-based virtual ligand screening.As Principal Investigator discussed before that (13cRA) is the strongest down-regulator of ACE2. and the principal investigator expects that 13cRA can inhibit or dowenrgulat ACE2 by direc interaction and binding with the transmembrane ACE2, Suggesting its therapeutic potential in preventing the entry of COVID 2019 to the host cell.

Previous studies on the related severe acute respiratory syndrome coronavirus (SARS-CoV) and SARS-CoV FP FP have shown that calcium (Ca2+) plays an important role for fusogenic activity via a Ca2+ binding pocket with conserved glutamic acid (E) and aspartic acid (D) residuesdemonstrated that intracellular Ca2+ enhances MERS-CoV WT PPs infection by approximately two-fold and that E891 is a crucial residue for Ca2+interaction. Electron spin resonance revealed that this enhancement could be attributed to Ca2+ increasing MERS-CoV FP fusion-relevant membrane ordering. Intriguingly, isothermal calorimetry titration showed that MERS-CoV FP binds one Ca2+, as opposed to SARS-CoV FP which binds to two Ca2+ ion.

Angiotensin II increases the intracellular calcium activity in podocytes of the intact glomerulus. The L-type Ca2+ channel blocker nicardipine did not influence the Ang II-mediated [Ca2+] increase and it has been postulated that SARS-CoV-2 binding to ACE2 may attenuate residual ACE2 activity, skewing the ACE/ACE2 balance to a state of heightened angiotensin II activity leading to pulmonary vasoconstriction and inflammatory and oxidative organ damage, which increases the risk for acute lung injury (ALI). AngII via AT1 receptors upregulates many proinflammatory genes, such as vascular cell adhesion molecule-1 (VCAM-1), intercellular adhesion molecule-1 (ICAM-1), interleukin-6 (IL-6).30 but 13cis RA specifically down-regulated the AT1 protein in a dose- and time-dependent manner. Down-regulation of the AT1 expression leads to reduced AngII-mediated intracellular calcium release Similarly with receptor down-regulation, Treatment with 13cRA resulted in a significant reduction in AT1 mRNA .13cRA has a glucose- and RAR/RXR independent mechanism for transcriptional inhibition of AT1,

Isotretinoin(13cis RA) may be able to inhibit COVID 2019 infection via reversIing the androgenic induction and activation effect of (DHT) on TMPRSS2 expression and helps to prevent cleaving and activating both the spike protein (S) of COVID 2019 and the viral receptor, and this is discussed as follow :

TMPRSS2 is both the most frequently altered gene in primary prostate cancer and a critical factor enabling cellular infection by coronaviruses, including SARS-CoV-2. The modulation of its expression by steroids could contribute to the male predominance of severe infections and given that TMPRSS2 has no known indispensable functions, and inhibitors are available, it is an appealing target for prevention or treatment of respiratory viral infections

TMPRSS2, a key regulator in prostate cancerTMPRSS2 was first identified in prostate cancer shortly after the gene had been originally cloned. Prostate cancer cell lines strongly upregulated TMPRSS2 expression in response to androgens . TMPRSS2 is expressed on the luminal side of the prostate epithelium, and its expression is increased in prostate cancer tissue compared to non-cancerous prostate tissue. Notably, the TMPRSS2 gene is a partner in one of the most common gene fusion eventsin solid tumors: somatic gene rearrangements involving TMPRSS2 witha member of the ETS family of oncogenic transcription factors, most commonly ERG. This fusion occurs in approximately 50% of primary prostate cancers among men of European ancestry.While ERG is not normally regulated by androgen, the gene fusion juxtaposes the androgen receptor regulatory elements of TMPRSS2 with the ERG gene. The ERG gene is consequently controlled by androgen receptor signaling and expressed highly in prostate cancers harboring the TMPRSS2: ERG fusion. Intriguingly, the prevalence of the TMPRSS2: ERG fusion is lower in prostate tumors of both black and Asian men. The relevance of this to the current COVID-19 pandemic is unclear.TMPRSS2: ERG fusion- cancers also have a distinct set of risk factors related to hormonal signaling. For example, men with higher genetically determined transcriptional activity of the androgen receptor have a higher risk of TMPRSS2: ERG fusion-positive prostate cancer but not of fusion-negative prostate cancer

TMPRSS2 is an androgen receptor signaling target gene and an androgen-regulated cell-surface serine protease expressed predominantly in prostate and lung epithelial cell TMPRSS2 is normally expressed several fold higher in the prostate relative to any other human tissue, though the normal physiological function(s) remains unknown. Importantly, unlike other TTSPs, TMPRSS2 transcription is regulated by androgenic ligands and the androgen receptor (AR). There is a positive correlation between AR and TMPRSS2 in microdissected primary tumor epithelium (r2 = 0.39 ; p <0.001).

Dihydrotestosterone (DHT) significantly and dramatically induced the expression of TMPRSS2 protein with two molecular masses of 60 (full-length) and 38 kDa (N-terminus) in a dose responsive manner

Data from Chinese outbreak show death rates for men almost 50 per cent higher than for women show that Early research from China suggests women and children are less likely to die than men if they catch the coronavirus. Death rates for Covid-19, the disease those infected with the coronavirus develop, are low for everyone: only 2.4 per cent of the 44,672 people in the Chinese study died. But although roughly even numbers of men and women catch the disease, men are more likely to develop such a serious case of Covid-19 they die.

More than 70 percent of Italy's coronavirus deaths have been among men but scientists there admit they are mystified by the gender gap. At least 3,400 people in Italy have died of the devastating disease - it yesterday announced it had a higher death Toll than China - but less than 1,000 of them have been women. Men are also more likely to pick up the infection in the first place and account for 60 percent of confirmed cases, according to Italy's public health research agency. An earlier analysis found that 80 per cent of the deaths were in men and just 20 per cent were in women - but the gap has narrowed over time

According to this data the principal investigator thinks that there is a strong relation between high mortality in males and androgenic effect specifically the effect of DHT on TMPRSS2 protein which is used by covid 2019 in cell invasion and entry and depending on this data related to six hormones specifically (DHT) , The investigator was able to discover whey women and children less likely to die from illness than men. So, the investigator divided infected patients according to their six hormone because TMPRSS2 is an androgen-regulated cell-surface serine protease expressed predominantly in prostate and lung epithelial cell TMPRSS2.

Androgen(DHT) potential effect on TMPRSS2 expression in children is less than its effect in females and males followed by viral severity and vigrousity in men compared with children and women. .

Androgen (DHT) potential effect on TMPRSS2 expression in females is less than in males followed by viral severity and vigrousity in men compared with females .

So, the principal investigator thinks that when some researchers investigated the role of sex steroids in SARS-CoV pathogenesis by comparing gonadectomized and control counterparts after infection. Gonadectomy or treatment with flutamide, a non-steroidal anti-androgen did not affect morbidity and mortality in male mice following lethal MA15 infection, They may be were wrong in their conclusions in suggesting that androgens do not play a role in SARS-CoV pathogenesis because Gonadectomy or treatment with flutamide will not completely affect or inhibit DHT and its derivatives(5α-Androstan-3α,17β-Diol) concentration in tissues and blood because after inhibiting testosterone with flutamide . the pathway of DHT formation will be activated to compensate the inhibited testosterone levels so the TMPRSS2 expression will be significantly induced by DHT and the treated animals will not be affected in case of flutamide treatment but in case of Gonadectomy the expression of TMPRSS2 will be decreased by DHT inhibition only if along time has passed on Gonadectomy in order to make sure that DHT and its derivatives completely declined in levels that will not allow it to affect on expression of TMPRSS2 and in female mice after blocking estrogen receptors it died because increasing formation of androgenic hormones.

A study demonstrated that 13- cis -Retinoic acid competitively and reversibly inhibits Dihydrotestosterone So, the principal investigator expects a significant modulation of TMPRSS2 expression after treating with 13- cis -Retinoic acid via temporary preventing the effect of dihydrotestosterone(DHT) on TMPRSS2 promoting and expression. And the type II transmembrane serine proteases TMPRSS2 which can cleave and activate the spike protein (S) of the severe acute respiratory syndrome coronavirus (SARS-CoV) for membrane fusion. In addition, these proteases cleave the viral receptor, the carboxypeptidase angiotensin-converting enzyme 2 (ACE2), and it was proposed that ACE2 cleavage augments viral infectivity.

A study demonstrated that COVID-19 reduces testosterone levels in men by altering the functioning of the gonads. So could the increased severity of the disease in men be due to lowered testosterone. But according to the principal investigator explanation COVID-19 reduces testosterone levels because there is a dramatic reductions in the cholesterol levels of patients infected with COVID 19, compared with healthy controls . Cholesterol levels decline quite rapidly during the early stages of infection and increase as the patient starts to recover.Therefore, indicating that cholesterol may have an important role to play in defending the body against such infections and depending on the principal investigator explanation, Testosterone is synthesized starting from cholesterol through a well-characterized steroid biosynthetic pathway involving the sequential action of multiple enzymes So, when cholesterol levels are decreased, this decrease will followed by decreasing in testosterone level and according to this explanation testosterone therapy in COVID 2019 is not recommended but temporary inhibitor of DHT is recommended such as Isotretinoin because this treatment by testosterone will inhibit cholesterol synthesis by feedback inhibition and decrease cholesterol uptake by Leydig cells in testis and this also will lead to over increase in DHT lvels and its derivatives in different tissues, which will induce TMPRSS2. because DHT is a potent activator of TMPRSS2 and this will be followed by processing and activation of COVID2019 spike protein to bined its ACE2 receptors in lung and kidney leading to their damage specifically in testis because it contains high levels of proteases and ACE2. Serine proteases are emerging as important contributors to the production, maturation, and functional competence of spermatozoa.

Tamoxifen may be able to inhibit COVID 2019 by inhibition acidification of the endosomes and lysosomes rather than inhibition of lysosomal enzymes.

A study demonstrated that tamoxifen causes redistribution of weak base chemotherapeutics from acidic organelles to the nucleus in drug-resistant cells. Agents that disrupt organelle acidification (e.g., monensin, bafilomycin A1) cause a similar redistribution. Measurement of cellular pH in several cell lines reveals that tamoxifen inhibits acidification of endosomes and lysosomes without affecting cytoplasmic pH. Similar to monensin, tamoxifen decreased the rate of vesicular transport though the recycling and secretory pathways. Organellar acidification is required for many cellular functions, and its disruption could account for many of the side effects of tamoxifen. A sudy demonstrated that the phagocytosis is inhabited by tamoxifen and chloroquine in retinal epithelial cells A study demonstrated that Tamoxifen have weak base property and increase endolysosomal pH and alter endosomal dynamics. Importantly, TAM treatment enhanced survival of mice injected with a lethal dose of STx1 or STx2,The protective effect was independent of estrogen receptors but dependent on the weak base property of TAM, which allowed TAM to increase endolysosomal pH and alter endosomal dynamics. A study demonstrated that Tamoxifen have antimalarial effect via treating mice infected with P. berghei, which show lower levels of parasitaemia and do not develop signs of cerebral malaria, Tamoxifen is found to prevent lung fibrosis and reduce serum TGFβ-1 levels. Astudy demonstrated that Tamoxifen have endosomal and lysosomal cysteine proteases inhibitory effect better than chloroquine , Cathepsins are endosomal and lysosomal cysteine proteases that play important roles in protein degradation in various cellular processes including both the endocytic pathway and autophagy. The role of cathepsins in viral infection was first identified by Huang et al and they found that one cysteine proteases inhibitor E64d and a specific cathepsin L inhibitor Z-FY(t-Bu)-DMK are able to block the SARS-CoV infection. Cathepsin D was more sensitive to tamoxifen than to chloroquine. Tamoxifen exposures decreased the cathepsin D activity at less than 10 pM concentrations. The effect of chloroquine started at 15 pM

.

ELIGIBILITY:
Inclusion Criteria:

Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

Age < 18 Pregnant Allergic to experimental drugs and patients have the following conditions:

1. Hypercholesterolemia
2. Hypertriglyceridemia
3. Liver disease
4. Renal disease
5. Sjögren syndrome
6. Pregnancy
7. Lactation
8. Depressive disorder
9. Body mass index less than 18 points or higher than 25 points
10. Contraindications for hormonal contraception or intrauterine device.
11. Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
12. Patients receiving anti-hcv treatment
13. Permanent blindness in one eye
14. History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery
15. The competent physician considered it inappropriate to participate in the study
16. bleeding dyscrasia

    16-1-anti-coagulation use active cervicitis
17. allergy to tamoxifen
18. history of venous thromboembolism
19. personal history of breast or uterine malignancy
20. use of medication contraindicated with use of tamoxifen (coumadin, letrozole, bromocriptine, rifampicin, aminoglutethimide, phenobarbital)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
lung injury score | at 7 days
  Proportion of lung injury score decreased or increased after treatment

SECONDARY OUTCOMES:
Absolute lymphocyte counts | at day 7 and 14
  lymphocyte counts
Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferon | at day 7 and 14
  Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferon
Serum level of COVID19 RNA | at day 7 and 14
  Serum level of COVID19 RNA
All cause mortality rate | at day 7 and 14
Ventilation free days | at 14 days
ICU free days | at 14 days
d-dimers | at 3-5 days
  less than 250 ng/mL, or less than 0.4 mcg/mL of blood sample
Time to first negative SARS-CoV-2 PCR in NP swap | 14 days
  (if pos. at baseline)